CLINICAL TRIAL: NCT00566605
Title: Visual Outcomes in a Comparison of Manual Penetrating Keratoplasty and the IntraLase® Enabled Keratoplasty
Brief Title: Outcomes in a Comparison of Manual Penetrating Keratoplasty and the IntraLase® Enabled Keratoplasty
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Oftalmologico de Sorocaba (Other)
Responsible Party: Luciene Barbosa de Sousa, HOSBOS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 466.07
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2007-12-03 (Estimated); Status verified 2007-11

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Keratoplasty, Penetrating

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Procedure: Penetrating keratoplasty with IntraLase
- Group 2 (Active Comparator)
  Interventions: Procedure: Penetrating keratoplasty with vacuum trephine

INTERVENTIONS:
Procedure: Penetrating keratoplasty with IntraLase — penetrating keratoplasty with femtosecond laser shaped incisions- IntraLase TM (IntraLase Enabled Keratoplasty [IEK])
  Arms: Group 1
Procedure: Penetrating keratoplasty with vacuum trephine — Group 2 - penetrating keratoplasty with vacuum trephine
  Arms: Group 2

SUMMARY:
To compare the early visual results and postoperative recovery between two groups of keratoconic patients - one group having undergone a traditional, mechanical vacuum trephine procedure while the second group underwent femtosecond-enabled penetrating keratoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old, with keratoconus and corneal transplant indication

Exclusion Criteria:

* Exclusion criteria included different ocular pathology and a potential visual acuity of less than 20/40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-08; Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 1 year

SECONDARY OUTCOMES:
Pachimetry, Microscopy, Corneal topography | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elissandro M Silva, Lindoso, Principal Investigator — Hospital Oftalmologico de Sorocaba
Locations (1):
- Sorocaba Eye Bank - HOSBOS, Sorocaba, São Paulo, Brazil